CLINICAL TRIAL: NCT05792852
Title: Feasibility of ENGAGE to Address Social Isolation Related to the COVID-19 Pandemic
Brief Title: Improving the Health and Social Participation of People With Disabilities From Underrepresented Groups Post COVID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Joy M Hammel, Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1393; UL1TR002003 (NIH)
Record Dates: First submitted 2023-03-27; First posted 2023-03-31 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Disabilities Multiple
MeSH Terms: interventions — engage 8200

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ENGAGE (Experimental): ENGAGE uses social learning, guided problem-solving and applied skill training to promote social participation among people with disabilities within the context of the COVID-19 pandemic. This is a group intervention using a self-management framework.
  Interventions: Behavioral: ENGAGE

INTERVENTIONS:
Behavioral: ENGAGE — ENGAGE is a group intervention designed to improve social participation within the context of the COVID-19 pandemic.

SUMMARY:
This is a single-arm community-based feasibility study examining recruitment, retention, adherence, and satisfaction with ENGAGE, a community-based intervention designed to address pandemic-related social isolation among people with disabilities. We will also examine preliminary, within-group effects on social participation. The findings of this study will inform a larger trial to examine intervention efficacy.

DETAILED DESCRIPTION:
Social isolation has been shown to negatively affect physical and mental health, particularly among people with disabilities. Social isolation among people with disabilities has been exacerbated by the COVID-19 pandemic. Even now, people with disabilities remain hesitant to return to social and community activities due to ongoing risk of severe cases and death. Yet, we do not have strong models of intervention designed to address this problem.

ENGAGE is an intervention that may address this gap. ENGAGE was designed to address social and community participation among people with stroke. We have since conducted qualitative research to inform adaptation of ENGAGE to meet the needs of a broader range of people with disabilities related to participation in the context of the ongoing COVID-19 pandemic. This study is the next step in testing and refining the adapted intervention protocol. At the end of this study, we will have a finalized adapted intervention protocol ready for large-scale efficacy testing.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as disabled
* Report problems with social participation
* Speak English
* Live in a community setting

Exclusion Criteria:

* Severe communication impairment limiting ability to verbally indicate interest in participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | 8 weeks
  Recruitment (5-7 participants per group recruited within one month), retention (80% of participants complete follow up assessments), adherence (80% of participants complete the intervention group
Intervention Satisfaction | 8 weeks
  Client Satisfaction Questionnaire-8: 8-item scale of intervention satisfaction with a 32-point scale (higher scores indicate greater satisfaction). We will establish adequate acceptability if we achieve a mean score of 24 or greater.

SECONDARY OUTCOMES:
Social Participation | 8 weeks
  PROMIS Ability to Participate in Social Roles (Cohen's d=/> .2)

CONTACTS AND LOCATIONS:
Overall Officials: Joy Hammel, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No